CLINICAL TRIAL: NCT06272448
Title: teleRehabilitation for pAtients With ParkInson's Disease at Any mOment
Acronym: RAPIDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Politecnica delle Marche (Other)
Collaborators: Universita di Verona (Other)
Responsible Party: Principal Investigator, Marianna Capecci, PhD, Prof., Università Politecnica delle Marche
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERM2022-27 21042022
Record Dates: First submitted 2023-01-16; First posted 2024-02-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
Keywords: Telerehabilitation; Telemonitoring; Empowerment; Functioning
MeSH Terms: conditions — Parkinson Disease; Empowerment | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Before-after study with one follow-up at 3 months of treatment end
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Telerehabilitation for 3 months
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — The subjects will be instructed to login with own credentials to a telerehabilitation platform where a library of videoclips displaying as many different motor activities, grouped by difficulty and function domain (trunk alignment, balance, hand dexterity, speech articulation, ventilation…), will be available. Patients will perform the exercises, according to a pre-determined training protocol, observing and imitating the tasks presented by the videoclips, for a total 45 minutes/day, at least 3 times/week (for no less than 27 sessions in total, equal to 1200 minutes of training). Subjects will be given a smartwatch to be worn 24 hours/ day, for at least 5 days/week. Every 15 +/- 3 days, one physiotherapist will call the patients to check the correct use of the devices, the level of adherence to the exercise program and the need for shaping the training difficulty to the user's skills

SUMMARY:
The goal of this clinical trial is to test the feasibility and safety of a telerehabilitation and telemonitoring approach in people with Parkinson's disease at any stage. The main questions it aims to answer are: will patients with Parkinson's disease comply with the recommended level of training at home using an ad hoc developed telerehabilitation platform? • Will this training be safe and impact the patient's well-being perception? Participants will be given a tablet and instructed to access an online platform to observe different motor tasks presented in as many video clips by experienced therapists.They will be requested to perform the motor tasks per a predetermined protocol over 3 months. Their compliance with the recommended training will be checked by physiotherapists every 15 days during phone calls, whereas their daily level of motor activity will be recorded by a smartwatch.

DETAILED DESCRIPTION:
In this cohort study, the feasibility and safety of a telerehabilitation and telemonitoring approach will be tested in people with Parkinson's disease at any stage. Enrolled subjects will be given a tablet through which they will log in with their own credentials to a telerehabilitation platform where a library of videoclips displaying as many different motor activities, grouped by difficulty (very easy - easy- advanced) and function domain (trunk alignment, balance, hand dexterity, speech articulation, ventilation…), will be available. Patients will perform the exercises according to a pre-determined training protocol, observing and imitating the tasks presented in the videoclips by experienced physiotherapists or speech therapists. A training duration of 45 minutes/day, 3 times/week for no less than 27 sessions (equal to 1200 minutes of total training) will be recommended. Moreover, subjects will be given a smartwatch to be worn 24 hours/ day, for at least 5 days/week. Every 15 +/- 3 days, one physiotherapist will call the patients to check the correct use of the devices, the level of adherence to the exercise program and the need for shaping the training difficulty to the user's skills.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease (according to Movement Disorder Society criteria)
* Ability to provide written informed consent.

Exclusion Criteria:

* moderate-severe cognitive impairment (MoCA≤18)
* any other factor known to interfere with the ability to interact with the telerehabilitation platform (e.g. poor visual acuity, lack of family support);
* comorbidities with adverse impact on functioning or survival or affecting the performance of physical exercise (e.g. serious neoplastic diseases, cardiovascular diseases not controlled pharmacologically including arterial hypertension or hypotension, cardiac arrhythmias, heart failure, musculoskeletal diseases, dizziness or vertigo);
* severe depression or other neuropsychiatric disorders;
* expected need for adapting antiparkinsonian drug regimen over a 6 month period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Compliance with the telerehabilitation system | At 3 months of baseline (end of treatment)
  Number of training sessions / minimum number of recommended sessions (i.e. at least 27 sessions) over 3 months
Perceived usability of system | At 3 months of baseline (end of treatment)
  SYSTEM USABILITY SCALE (range 0-100, with 100 being the maximum usability perception)
Incidence of treatment-emergent adverse events | At 3 months of baseline (end of treatment)
  N. of adverse events occurring while using the telerehabilitation system

SECONDARY OUTCOMES:
User satisfaction | At 3 months of baseline (end of treatment)
  Patient Global Rating of Change (range: from -3 to + 3, with negative scores conveying a perception of worsening)
Compliance with the monitoring system | At 3 months of baseline (end of treatment)
  Total smartwatch activation duration/minimum expected activation duration (i.e. 24 hours/day x 3 months)
Feasibility of telemonitoring approach | At 3 months of baseline (end of treatment)
  (n. of remote contacts with the physiotherapists/minimum number of planned contacts (i.e. at least 5 over 3 months);
Motor symptom and disability progression | At baseline and 3 and 6 months after
  Change in the Unified Parkinson's Disease Rating Scale score (range 0-260, 0= no symptoms, complete independence)
Non motor symptom progression | At baseline and 3 and 6 months after
  Change in the NonMotor Symptoms Scale score (range 0-360, 0= no symptoms)
Patients' Quality of life | At baseline and 3 and 6 months after
  Change in Parkinson's Disease Questionnaire PDQ-8 score (range 0-32, 0=best quality of life)
Caregiver's burden | At baseline and 3 and 6 months after
  Change in ZARIT BURDEN INTERVIEW 22.item score (range 0-88, 0= best condition)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gabriella Ceravolo, Prof, Principal Investigator — Politecnica delle Marche University
Locations (2):
- Italy (2):
  - Neurorehabilitation Clinic, Ancona
  - Università di Verona, Verona